CLINICAL TRIAL: NCT02847689
Title: Listening to Mom in the Neonatal Intensive Care Unit (NICU): Neural, Clinical and Language Outcomes
Brief Title: Listening to Mom in the NICU: Neural, Clinical and Language Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Katherine E Travis, PhD, Instructor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 32638; 1K99HD084749-01A1 (NIH)
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Premature Birth
Keywords: Premature Birth; Obstetric Labor, Premature; Obstetric Labor Complications; Pregnancy Complications
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Obstetric Labor Complications; Pregnancy Complications | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Language Treatment Arm (Experimental): An infant participant randomized to the language treatment arm will be played recordings of his/her mother's voice 2-3 hours daily in the intermediate care nursery until discharge.
  Interventions: Behavioral: Language Treatment
- Control Treatment Arm (Sham Comparator): An infant participant randomized to the control treatment arm will receive standard of care. Standard of care does not include being played recordings of his/her mother's voice while admitted to the intermediate care nursery. However, an infant randomized to the control treatment will have the same auditory equipment placed in his/her isolette or crib as an infant randomized to the Language Treatment Arm.
  Interventions: Behavioral: Control Treatment

INTERVENTIONS:
Behavioral: Language Treatment — Recording of a mother's voice reading a children's storybook.
  Arms: Language Treatment Arm
Behavioral: Control Treatment — Standard of Care
  Other Names: Standard of Care
  Arms: Control Treatment Arm

SUMMARY:
The purpose of this study is to examine whether playing recordings of a mother's voice to her infant while in the hospital nursery is an effective treatment for promoting healthy brain and language development in infants born preterm.

DETAILED DESCRIPTION:
Children born preterm are at-risk for developmental language delays. Language problems in preterm children are thought to be related to neurobiological factors, including injuries to white matter structures of the brain and environmental factors, including decreased exposure to maternal speech in the hospital nursery. There is evidence to suggest that maternal speech input may be important for promoting healthy brain and language development.

Participants will be randomly assigned to one of two study groups. Each infant has a 50% chance of being assigned to the group that will listen to a recording of his/her mother's voice and a 50% chance of being assigned to the group that will not be played a voice recording. Mother's of participating infants will have her voice recorded as she reads a common children's storybook. Recordings will be played to infants each day until s/he is discharged from the hospital. Participation in this study requires that all infants receive up to an additional 10 minutes of brain scans as part of his/her routine clinical magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Infants born preterm at Stanford Children's Hospital between 27 0/7 - 31 6/7 weeks gestational age

Exclusion Criteria:

* Congenital anomalies
* Recognizable malformation syndromes
* Active seizure disorders
* History of Central Nervous System infections
* Hydrocephalus
* Major sensori-neural hearing loss
* Likelihood to be transferred from NICU to alternate care facility or home environment prior to 36 weeks PMA
* Intraventricular Hemorrhage Grades III-IV
* Cystic periventricular leukomalacia (PVL)
* Surgical treatment for necrotizing enterocolitis
* Small for gestational age (SGA) <3 percentile and/or Intra-uterine growth restriction (IUGR) no head sparing
* Twin-to-twin transfusions

Ages: 24 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2016-07; Primary Completion 2019-06-12 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
White matter mean diffusivity | 36-37 weeks post-menstrual age or at time of hospital discharge, whichever comes first
  Mean diffusivity measures the average rate of water diffusion within a given MRI voxel.

SECONDARY OUTCOMES:
Length of hospital stay | Days in hospital since birth and until discharge, average range is 37-40 weeks postmenstrual age (PMA)
  Days in hospital since birth and until discharge
Average daily weight gain | measured daily and beginning at start of treatment and until end of treatment, approximately 37-40 weeks PMA
Time (days) to full oral feed | measured daily and beginning at start of treatment and until end of treatment, approximately 37-40 weeks PMA
  days until 100 % of nutrition administered orally
Number of significant apnea and bradycardia events requiring stimulation | measured daily and beginning at start of treatment and until end of treatment, approximately 37-40 weeks PMA

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Travis, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University - Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT02847689/ICF_000.pdf